CLINICAL TRIAL: NCT02634827
Title: A Phase II Study of Combination Midostaurin and Decitabine (MIDDAC) in Elderly Patients Newly Diagnosed With Acute Myeloid Leukemia and FLT3 Mutation
Brief Title: Midostaurin and Decitabine in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia and FLT3 Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1483; NCI-2015-02107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1483 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2018-06

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation; Acute Myeloid Leukemia With Gene Mutations; FLT3 Tyrosine Kinase Domain Point Mutation; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: interventions — Decitabine; Injections; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (decitabine, midostaurin) (Experimental): Patients receive decitabine intravenously (IV) over 1 hour on days 1-5 and midostaurin orally (PO) twice daily (BID) on days 8-21 of courses 1 and 2, and on days 1-28 of each subsequent course. Patients failing to achieve complete response (CR)/complete response with incomplete recovery (CRi)/partial response (PR)/morphologic leukemia-free state by end of course 2 receive midostaurin PO BID on days 1-28. Patients achieving CR/CRi/PR/morphologic leukemia-free state by end of course 8 may continue on current regimen. Patients failing to achieve a CR/CRi/PR/ morphologic leukemia-free state in bone marrow blasts by end of course 8 go to event monitoring. Treatment repeats every 28 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis; Drug: Midostaurin

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Midostaurin — Given PO
  Other Names: CGP 41251; CGP41251; N-Benzoyl-Staurosporine; N-Benzoylstaurosporine; PKC-412; PKC412

SUMMARY:
This phase II trial studies how well midostaurin and decitabine work in treating older patients with newly diagnosed acute myeloid leukemia and FLT3 mutations. Midostaurin and decitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rate for elderly patients with FLT3 mutated acute myeloid leukemia (AML) using midostaurin and decitabine.

SECONDARY OBJECTIVES:

I. Determine the 1-year overall survival (OS) and progression free survival (PFS) rates.

II. Determine overall response rates in patients treated with this regimen. III. Determine the complete response duration in patients treated with this regimen.

IV. Assess the safety and toxicity of this regimen based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

TERTIARY OBJECTIVES:

I. Assess the prognostic and predictive factors (FLT3 internal tandem duplication [ITD] versus [vs] tyrosine kinase domain [TKD] mutation) for patients treated with this regimen.

II. Explore genetic targets for this disease.

OUTLINE:

Patients receive decitabine intravenously (IV) over 1 hour on days 1-5 and midostaurin orally (PO) twice daily (BID) on days 8-21 of courses 1 and 2, and on days 1-28 of each subsequent course. Patients failing to achieve complete response (CR)/complete response with incomplete recovery (CRi)/partial response (PR)/morphologic leukemia-free state by end of course 2 receive midostaurin PO BID on days 1-28. Patients achieving CR/CRi/PR/morphologic leukemia-free state by end of course 8 may continue on current regimen. Patients failing to achieve a CR/CRi/PR/ morphologic leukemia-free state in bone marrow blasts by end of course 8 go to event monitoring. Treatment repeats every 28 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Unfit for chemotherapy based on investigator assessment or patient not willing to receive intensive induction as advised by investigator
* Untreated, histological confirmed acute myeloid leukemia (AML) based on World Health Organization (WHO) 2008 criteria with either/or both:

  * FLT3 ITD mutation
  * FLT3 TKD mutation
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, 2 or 3
* Serum amylase and lipase =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN (does not apply to patients with isolated hyperbilirubinemia [e.g., Gilbert's disease], in that case direct bilirubin should be =< 2 x ULN)
* Alkaline phosphatase =< 3 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN
* Creatinine =< 2 x ULN
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to return to consenting Mayo Clinic (Mayo Clinic's campus in Rochester), for follow-up during the Active Monitoring Phase of the study
* Willing to provide bone marrow aspirate and blood samples for correlative research purposes

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after treatment completion
* Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject; NOTE: periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening); NOTE: for female subjects on the study the vasectomized male partner should be the sole partner for that subject
  * Combination of any two of the following (a+b or a+c, or b+c):

    * a) Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
    * b) Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * c) Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * NOTE:

    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment
    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) OR
  * Sexually active males unless they use a condom during intercourse while taking drug and for 5 months after stopping midostaurin medication
  * NOTE:

    * They should not father a child in this period
    * A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients confirmed to be human immunodeficiency virus (HIV) positive or have active viral hepatitis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements; patients with any other known concurrent severe and/or uncontrolled medical condition (except carcinoma in-situ), which could compromise participation in the study (e.g. uncontrolled infection, uncontrolled diabetes, chronic active pancreatitis)
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 1 year prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix
* Previous treatment with specific chemotherapy (cytarabine, idarubicin, daunorubicin) or hypomethylating drug (decitabine or azacitidine) for a hematological disorder; EXCEPTIONS: prior hydroxyurea allowed; secondary AML is allowed
* Impaired cardiac function including any of the following:

  * Inability to monitor the QT interval on electrocardiogram (ECG)
  * Congenital long QT syndrome or a known family history of long QT syndrome
  * Clinically significant resting brachycardia (< 50 beats per minute)
  * Corrected QT (QTc) > 450 msec on baseline ECG; NOTE: if the ECG shows a QTc interval greater than 450 msecs at screening triplicates should be performed, one minute apart to confirm the finding (after replacement of any electrolyte imbalance); if 2/3 or 3/3 of the ECGs confirm the QT prolongation (i.e. QTc interval > 450 msecs) the patient must not be included into the trial
  * Myocardial infarction =< 3 months prior to starting study
  * Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension)
  * History of or presence of clinically significant ventricular, atrial tachyarrhythmias or ejection fraction cutoff
  * Left ventricle ejection fraction < 45%
  * History of congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Patients currently receiving treatment with strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors and treatment that cannot be either discontinued or switched to a different medication prior to starting study drug; patients receiving any medications or substances that are strong inhibitors of CYP3A4; all azoles but fluconazole are discouraged to be used in patients requiring treatment with antifungal antibiotics; use of the following strong inhibitors is prohibited =< 7 days prior to registration

  * Strong inhibitors of CYP3A4/5; > 5-fold increase in the plasma area under the curve (AUC) values or more than 80% decrease in clearance

    * Boceprevir (Victrelis)
    * Clarithromycin (Biaxin, Biaxin XL)
    * Conivaptan (Vaprisol)
    * Indinavir (Crixivan)
    * Itraconazole (Sporanox)
    * Ketoconazole (Nizoral)
    * Lopinavir/Ritonavir (Kaletra)
    * Mibefradil
    * Nefazodone (Serzone)
    * Nelfinavir (Viracept)
    * Posaconazole (Noxafil)
    * Ritonavir (Novir®, Kaletra)
    * Saquinivir (Fortovase, Invirase)
    * Telaprevir (Incivek)
    * Telithromycin (Ketek)
    * Voriconazole (Vfend)
    * Troleandomycin
    * Cobicistat
    * Tipranavir
* Receiving any medications or substances that are inducers of CYP3A4; use of the following inducers are prohibited =< 7 days prior to registration

  * Strong inducers of CYP3A4/5; > 80% decrease in AUC

    * Avasimibe
    * Carbamazepine (Carbatrol, Epitol, Equetro, Tegretol, Tegretol-XR)
    * Phenytoin (Dilantin, Phenytek)
    * Rifampin (Rifadin)
    * St. John's wort
    * Mitotane
    * Rifabutin
    * Phenobarbital
  * Moderate inducers of CYP3A4/5; 50-80% decrease in AUC

    * Bosentan (Tracleer)
    * Efavirenz (Sustiva)
    * Etravirine (Intelence)
    * Modafinil (Provigil)
    * Nafcillin
    * Genistein
    * Ritonavir
    * Talyiraline
    * Thioridazine
    * Tipranavir
    * Nevirapine (Viramune)
    * Phenobarbital (Luminal)
    * Rifabutin (Mycobutin)
    * Troglitazone
* Patients currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug; NOTE: prohibited medications contains drugs that should be used with caution due to possible or conditional risk of Torsades de Pointes
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery)
* Acute or chronic pancreatic disease
* Known cytopathologically confirmed central nervous system (CNS) infiltration
* Acute or chronic liver disease or severe renal disease considered unrelated to the cancer
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Major surgery =< 4 weeks prior to registration of the study or who have not recovered from prior surgery regardless of time since surgery
* Treatment with other investigational agents =< 30 days or 5 half-lives of registration
* Diagnosis of AML-M3 (or acute promyelocytic leukemia)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2017-03-18 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aref Al-Kali, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One (1) patient was accrued from December 2015 to June 2018 at Mayo Clinic. Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Period: Overall Study
Arm/Group | Treatment (Decitabine, Midostaurin)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male
Race (NIH/OMB)
ECOG Performance Status

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Complete Responses to Therapy, Where a Success is Defined as a CR or CRi as the Objective Status
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial confidence intervals for the true success proportion will be calculated.
Time Frame: Up to 2 years
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Complete Response, Defined for All Evaluable Patients Who Have Achieved a CR or CRi as the Date at Which the Patient's Objective Status is First Noted to be a CR or CRi to the Earliest Date Relapse is Documented
Description: The distribution of duration of complete response will be estimated using the method of Kaplan-Meier. If there are a sufficient number of CR/CRi, a landmark analyses may be performed to compare duration of CR/CRi in patients who first achieved a CR/CRi at 2 months vs those who first achieved a CR/CRi at 8 months.
Time Frame: Up to 2 year
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Adverse Events, Graded According to the NCI CTCAE Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 2 years
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

4. Secondary Outcome: OS
Description: Estimated using the method of Kaplan-Meier. In addition, the overall survival rate at 1 year after registration will be reported.
Time Frame: Time from registration to death due to any cause, assessed up to 2 years
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Response Rate, Estimated by the Total Number of Complete or Partial Responses (CR, CRi, Morphologic Leukemia-free State, or PR) Divided by the Total Number of Evaluable Patients
Description: Overall response rate, estimated by the total number of complete or partial responses (CR, CRi, morphologic leukemia-free state, or PR) divided by the total number of evaluable patients Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Time Frame: Up to 2 years
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

6. Secondary Outcome: PFS
Description: Estimated using the method of Kaplan-Meier. In addition, the progression-free survival rate at 1 year after registration will be reported.
Time Frame: Time from registration to the time of relapse or death due to any cause, assessed up to 2 years
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: FLT3 Mutation by ITD vs. TKD vs. Both, Assessed by Polymerase Chain Reaction (PCR), Western Blot, and Flow Cytometry
Description: Prognostic and predictive factors including age and FLT3 mutation by ITD vs. TKD vs. both will be assessed. These factors will be summarized and used to help characterize the types of patients accrued to this trial. In addition, differences in the distributions of these risk factors by clinical outcome will be explored (CR/CRi vs. not, OS and disease-free survival). Nonparametric quantitative comparisons by group will be made as appropriate (Fisher's exact or Wilcoxon rank sum). Kaplan-Meier methods and log rank statistics will be used to compare between groups for time to- event measures.
Time Frame: Up to day 1 of course 9
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Minimal Residual Disease (MRD) Status, Assessed by PCR for FLT3 Mutation (if FLT3 is Repeated) or Flow Cytometry
Description: MRD status will be correlated with response using Fisher's exact test. In addition, the relationship between MRD status (positive vs. negative) and disease-free survival will be evaluated using landmark analyses.
Time Frame: Up to day 1 of course 9
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Treatment (Decitabine, Midostaurin)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT02634827/Prot_SAP_000.pdf